CLINICAL TRIAL: NCT05491213
Title: TELEhealth Shared Decision-making COaching for Lung Cancer Screening in Primary carE (TELESCOPE)
Brief Title: TELESCOPE- TELEhealth Shared Decision-making COaching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anita Y. Kinney, PhD, RN, Director at Rutgers Cancer Institute, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 132207; Pro2022000340 (Other: Rutgers); 1R01HL158850-01A1 (NIH)
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Lung Neoplasms
Keywords: Lung cancer screening; Shared decision making
MeSH Terms: conditions — Lung Neoplasms | interventions — Telescopes

STUDY DESIGN:
Intervention Model Description: Quantitative measures of the PRISM constructs will be collected via internet surveys from the patient and nurse navigators, clinic directors, and clinicians (n = 130 surveys), and through medical record review. Participants followed at the TELESCOPE arm sites will also complete a measure of intervention acceptability at the one week survey for Aim 2. Semi-structured interviews will be conducted for Aim 2 with a mix of 20 clinical, nursing, and administrative directors at the participating sites. All 10 study navigators, and 20 clinicians from the TELESCOPE arm sites will also be interviewed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TELESCOPE intervention (Experimental): Participants will be surveyed at baseline and at one-week after the scheduled primary care office visit. If a participant is a current smoker then they are offered and navigated to evidence-based smoking cessation. If the participant is interested in screening, an LDCT is ordered. Support for screening, diagnostic testing and oncology care will be provided as needed from the Nurse Navigators.
  Interventions: Behavioral: TELESCOPE, Remote Decision Coaching with Navigation Intervention
- Enhanced usual care (EUC) (No Intervention): Participants will be surveyed at baseline and at one-week after the scheduled primary care office visit. Primary and secondary outcome data related to the office visit will be collected.

INTERVENTIONS:
Behavioral: TELESCOPE, Remote Decision Coaching with Navigation Intervention — The TELESCOPE intervention involves three complementary components: 1) decision aid and coaching for LCS, 2) referral of current smokers to evidence-based smoking cessation services, and 3) for participants interested in screening, navigation to complete LCS and diagnostic testing and oncology care as needed
  Arms: TELESCOPE intervention

SUMMARY:
Hypothesis 1a: The investigators anticipate that navigator decision coaching, compared to enhanced usual care (EUC) will result in higher quality SDM for lung cancer screening (LCS )(primary outcome), greater knowledge of lung cancer screening benefits and harms, and lower decisional conflict.

Hypothesis 1b: Compared to enhanced usual care (EUC), we expect that TELESCOPE will result in more screening discussions, increased initial for lung cancer screening (LCS) with low-dose CT scan (LDCT) uptake among interested participants, increased adherence to repeat LCS and diagnostic testing, and increased smoking cessation referrals for current smokers.

Hypothesis 2: The investigators expect that a "booster" coaching session will increase adherence to repeat lung cancer screening (LCS).

DETAILED DESCRIPTION:
The investigators' primary objective is to compare the effectiveness of the TELESCOPE intervention vs. enhanced usual care (EUC) on shared decision-making (SDM) for lung cancer screening.

Secondary objectives are to test the effectiveness of the TELESCOPE intervention vs. EUC on screening uptake, adherence with diagnostic testing and annual testing, and smoking cessation referrals and receipt of tobacco treatment for current smokers. The investigators will also use a mixed methods approach to evaluate the implementation potential of navigator-led decision coaching for lung cancer screening (LCS ) and identify components and organizational and individual level characteristics that might facilitate or interfere with successful implementation.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria Cluster Randomized Trial

Eligibility of patients for the cluster randomized trial will follow United States Preventive Services Task Force criteria for lung cancer screening. Specifically, patients must:

* Be 50 to 77 years of age
* Be a current or former smoker having quit within the past 15 years
* Have at least a 20 pack-year smoking history
* Be scheduled for a non-acute care visit at one of the study sites. Interviews (N=50)

Participants completing the semi-structured interviews will be:

* A practicing primary care clinician or a clinic director (n=20), nursing director, or clinic practice administrator (n=20) at one of the participating sites or a TELESCOPE study patient navigator (n=7) and nurse navigator (n = 3)
* Age 18 or older
* Fluent in English Online surveys (N=130)

Providers completing online PRISM construct surveys will be:

* A practicing primary care provider at one of the participating sites or a TELESCOPE study navigator
* Age 18 or older
* Fluent in English

Exclusion Criteria:

- Cluster Randomized Trial

Excluded will be patients who:

* Do not speak English
* Have a history lung cancer
* Were screened for lung cancer within the past 12 months
* Have health conditions that make them poor candidates for curative treatment as determined by the primary care provider
* Are unable to provide informed consent Interviews (N=50)

Providers/administrators will be excluded if they:

* Are unable to provide informed consent Online surveys (N=130)
* Are unable to provide informed consent
* Women who are pregnant. English proficiency is required for the completion of surveys, and the intervention will be conducted in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 594 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To assess shared decision making | The change in baseline, three months and five years
  Semi-structured interviews (qualitative data)

SECONDARY OUTCOMES:
Tobacco treatment referral | The change in baseline, three months and five years
  Semi-structured interviews (qualitative data)
Uptake of Low-Dose CT Screening for Lung Cancer | Within 6 months post-intervention
  Proportion of participants who complete low-dose CT (LDCT) lung cancer screening within 6 months post-intervention.

OTHER OUTCOMES:
Receipt of tobacco treatment | The change in baseline, three months and five years
  Semi-structured interviews (qualitative data).
Completion of diagnostic testing | The change in baseline, three months and five years
  Semi-structured interviews (qualitative data).

CONTACTS AND LOCATIONS:
Overall Officials: Anita Y Kinney, PhD, RN, Principal Investigator — Rutgers Cancer Institute
Locations (2):
- United States (2):
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan NQP, Lowenstein LM, Douglas EE, Silva J, Bershad JM, An J, Shete SS, Steinberg MB, Ferrante JM, Clark EC, Natale-Pereira A, Sahu NN, Hastings SE, Hoffman RM, Volk RJ, Kinney AY. The TELEhealth Shared decision-making COaching and navigation in Primary carE (TELESCOPE) intervention: a study protocol for delivering shared decision-making for lung cancer screening by patient navigators. BMC Prim Care. 2024 Oct 18;25(1):373. doi: 10.1186/s12875-024-02610-2. PMID 39425032
- [Derived] Tan NQP, Lowenstein LM, Douglas EE, Silva J, Bershad JM, An J, Shete SS, Steinberg MB, Ferrante JM, Clark EC, Natale-Pereira A, Sahu NN, Hastings SE, Hoffman RM, Volk RJ, Kinney AY. The TELEhealth Shared decision-making Coaching and Navigation in Primary carE (TELESCOPE) intervention: a study protocol for delivering shared decision-making for lung cancer screening by patient navigators. Res Sq [Preprint]. 2024 Apr 22:rs.3.rs-4254047. doi: 10.21203/rs.3.rs-4254047/v1. PMID 38746205